CLINICAL TRIAL: NCT01621022
Title: Efficacy of Bupropion Alone and in Combination With Nicotine Gum
Brief Title: Bupropion Alone or Combined With Nicotine Gum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB S-01-07
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Tobacco Dependence
Keywords: smoking cessation; tobacco dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Bupropion; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active bupropion-Active gum (Active Comparator): 150 mg bupropion twice daily + 4 mg nicotine gum as needed (up to 12 pcs/day)
  Interventions: Drug: bupropion + nicotine gum
- Active bupropion-Placebo gum (Active Comparator): 150mg bupropion twice daily + placebo gum as needed (up to 12 pcs/day)
  Interventions: Drug: Active bupropion-Placebo gum
- Placebo medication-Placebo gum (Active Comparator): Placebo bupropion, twice daily, plus placebo gum as needed (up to 12 pcs/day)
  Interventions: Drug: Placebo bupropion-Placebo gum

INTERVENTIONS:
Drug: bupropion + nicotine gum — 150 mg bupropion twice daily plus 4 mg nicotine gum as needed (up to 12 pcs/day)
  Arms: Active bupropion-Active gum
Drug: Active bupropion-Placebo gum — 150mg bupropion twice daily plus placebo nicotine gum as needed (up to 12 pcs/day)
  Arms: Active bupropion-Placebo gum
Drug: Placebo bupropion-Placebo gum — Placebo bupropion twice daily + placebo nicotine gum as needed (up to 12 pcs/day)
  Arms: Placebo medication-Placebo gum

SUMMARY:
Focus of this study was to determine if bupropion was more effective for smoking cessation when used alone or combined with nicotine gum.

ELIGIBILITY:
Inclusion Criteria:

* Smoke 10 or more cigarettes per day
* Motivated to quit
* No physical or mental health issues that would prevent participation
* Not pregnant or willing to prevent pregnancy during treatment

Exclusion Criteria:

* Carbon monoxide (CO) breath test score below 10 parts per million (ppm)
* Center for Epidemiologic Studies Depression Scale (CES-D) score greater than 16
* Heavy alcohol use
* History of eating disorder
* Suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2001-01; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence measured at 6 months | 6 months
  No smoking, not evan a puff, during the 7 days prior to the 6 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- UW Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

REFERENCES:
- [Result] Piper ME, Federman EB, McCarthy DE, Bolt DM, Smith SS, Fiore MC, Baker TB. Efficacy of bupropion alone and in combination with nicotine gum. Nicotine Tob Res. 2007 Sep;9(9):947-54. doi: 10.1080/14622200701540820. PMID 17763111
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961